CLINICAL TRIAL: NCT05087251
Title: Randomized Trial of an Intervention to Enhance Quality of Life in Adults Completing Lung Cancer Treatment With Curative Intent
Brief Title: The Transitions Project: Efficacy Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: American Lung Association (Other)
Responsible Party: Principal Investigator, Lara Traeger, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-426
Record Dates: First submitted 2021-10-01; First posted 2021-10-21 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; Supportive Care
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Five Psycho-educational Sessions (Experimental): Approximately 6 weeks after the patient's cancer treatment is complete, participants in the intervention arm will proceed to receive up to 5 study sessions (approximately weekly, ~50 minutes each) with a trained interventionist focused on psychoeducational topics. This arm was designed to enhance patient skills to address key concerns during the transition from treatment to surveillance, using a cognitive-behavioral approach. Sessions will be based on an intervention manual.
  Interventions: Behavioral: Five Psycho-educational Session(s)
- Enhanced Usual Care: One Psycho-educational Session (Experimental): At approximately 6 weeks after treatment completion (as defined by our eligibility criteria), control patients will attend one study session (~50 minutes) with a study clinician. This session is designed to control for patient access and connection to psychosocial resources as recommended in recent work.
  Interventions: Behavioral: One Psycho-educational Session(s)

INTERVENTIONS:
Behavioral: Five Psycho-educational Session(s) — 5 psychoeducational sessions focused on skills for enhancing wellbeing, relationships, social support, and ability to cope with uncertainty
  Arms: Intervention: Five Psycho-educational Sessions
Behavioral: One Psycho-educational Session(s) — 1 session focused on exploring goals and expectations for post-treatment quality of life, including supportive listening; assessment of unmet needs; preferences for support, and tailored referral recommendations
  Arms: Enhanced Usual Care: One Psycho-educational Session

SUMMARY:
The aim of this study is to evaluate the efficacy of a brief psychoeducational intervention to improve quality of life in patients with lung cancer who are transitioning from active treatment to surveillance.

DETAILED DESCRIPTION:
This is a randomized controlled trial to test the efficacy of a brief psychoeducational intervention relative to a control condition for improving quality of life in patients with lung cancer who are transitioning from treatment to surveillance.

In this study, participants will complete survey questions and will be randomly assigned to receive a 5-session program or a 1-session program.

It is expected that about 100 people will take part in this research study.

The American Lung Association is supporting this research by providing funding for the research study.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 or older
* Able to read and respond in English
* Diagnosis of non-small cell lung cancer or small cell lung cancer
* Documented curative treatment plan including systemic therapy +/- radiation and +/- surgery
* Completed cancer treatment within past 3 weeks

  * If final treatment is systemic therapy +/- radiation: within 3 weeks after cancer care team determination that treatment is complete
  * If final treatment is surgery: within 3 weeks after hospital discharge following surgery

Exclusion Criteria:

* Comorbid health condition that would interfere with study participation
* Current participation in cognitive behavioral therapy treatment

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Quality of life: Functional Assessment of Cancer Therapy-Lung Cancer | Up to 12 weeks
  We will investigate longitudinal differences in quality of life between study groups (Functional Assessment of Cancer Therapy-Lung Cancer score range 0-144, with higher scores indicating better quality of life)

SECONDARY OUTCOMES:
Fear of cancer recurrence: Fear of Cancer Recurrence Scale 7 | Up to 12 weeks
  We will investigate longitudinal differences in fear of cancer recurrence between study groups (Fear of Cancer Recurrence Scale 7, score range 7-35, with higher scores indicating more fear of cancer recurrence)
Symptom burden: Edmonton Symptom Assessment Scale | Up to 12 weeks
  We will investigate longitudinal differences in symptom burden (Edmonton Symptom Assessment Scale score range 0-90, with higher scores indicating more symptom burden)
Psychological symptom burden: Hospital Anxiety and Depression Scale | Up to 12 weeks
  We will investigate longitudinal differences in psychological symptom burden (Hospital Anxiety and Depression Scale score range 0-42 with higher scores indicating more psychological symptom burden)
Social support: Multidimensional Scale of Perceived Social Support | Up to 12 weeks
  We will investigate longitudinal differencs in social support (Multidimensional Scale of Perceived Social Support score range 12-84, with higher scores indicating more social support)
Social isolaton: Campaign to End Loneliness Measurement Tool | Up to 12 weeks
  We will investigate longitudinal differences in social isolation (Campaign to End Loneliness measurement tool score range 0-12 with higher scores indicating more social isolation)

CONTACTS AND LOCATIONS:
Overall Officials: Lara Traeger, PhD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation